CLINICAL TRIAL: NCT06734728
Title: Post-marketing Study for the Evaluation of the Efficacy and Safety of Profilm Cold Sores
Brief Title: Post-marketing Study for the Evaluation of Profilm Cold Sores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Dr. Goya Análisis, SL. (Industry); Centro Médico Complutense Grupo Virtus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROFILM HERPES-PIC01-2022
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cold Sores
Keywords: Herpes; Oral herpes simplex; Oral ulcer
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex; Stomatitis, Herpetic; Oral Ulcer

STUDY DESIGN:
Intervention Model Description: Intrasubject control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Profilm Cold Sores (Experimental): Participants will use Profil Cold Sores daily as soon as the first symptoms of a new outbreak appear and until the outbreak is resolved.
  Interventions: Device: Profilm Cold Sores

INTERVENTIONS:
Device: Profilm Cold Sores — The treatment will consist of daily applications of the product as soon as the first symptoms of an outbreak appear, and until the outbreak subsides, as follows: application every 8 hours, with the possibility of shortening the interval to 6 hours if needed (a maximum of 3-4 applications).

SUMMARY:
Experimental clinical study with a post-marketing, prospective, intra-subject controlled design to evaluate the efficacy and safety of the use of a medical device for the treatment of cold sores, over a maximum period of two weeks (or until the outbreak has resolved).

ELIGIBILITY:
nclusion Criteria:

* Male / female / aged 18 years or older.
* Presence of a herpes labial outbreak, regardless of the number of days since its appearance.
* At least 30 days have passed since the last episode.
* Willingness to return for all study-related visits.
* Sufficient willingness and ability, as judged by the investigator, to respond to the questionnaires included in the study.

Exclusion Criteria:

* Pregnant women or women in the breastfeeding period.
* Patients undergoing treatment with antiviral medications, hydrocortisone, or other medications.
* Patients with immunodeficiency diseases, such as acquired immunodeficiency syndrome or altered immune activity in the last 7 days.
* Patients undergoing other pharmacological therapy forrecurrent herpes labial.
* Patients with other oral mucosa diseases simultaneously.
* Known allergy or hypersensitivity to any of the components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Confirm the effectiveness of the treatment in terms of pain relief, using an EVA scale. | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  Pain relief as a significant clinical improvement in the EVA Pain score from 0 to 10 (where 0 = no pain and 10 = unbearable or severe pain) after treatment.
Serious adverse events. | Through study completion, apprroximately 2 weeks.
  Evaluate the safety of the treatment related to the product, in terms of the incidence of serious adverse events during the treatment.

SECONDARY OUTCOMES:
Evaluation of the treatment based on lesion size. | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  A decrease of at least 50% of the maximum size reached, at the midpoint of the treatment (7 days). Exploratory analysis at 14 days or at the end of the outbreak, with at least an 80% reduction in the extent of the lesion

OTHER OUTCOMES:
Changes in the intensity and severity of the symptoms. | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  Assessment of the severity-intensity of symptoms (pain, itching, burning or stinging, and tingling) perceived with a score ≤ 4 points on a 0 to 10 scale. (Where 0 = no symptoms / 10 = severe symptoms).
Degree of protection-hygiene provided by the treatment. | At the conclusion of the study, approximately 2 weeks later.
  It is done using a scale from 0 to 10, where 0 = no protection and 10 = full protection. A score of ≥ 5 on a scale from 0 to 10 at the end of the treatment will indicate effectiveness.
Evaluation of the visibility-noticeability of the outbreak. | At the conclusion of the study, approximately 2 weeks later.
  It will be done using a scale where a score of ≤ 5 on a scale from 0 to 10 at the end of the treatment will indicate effectiveness (where 0 = not noticeable at all and 10 = highly noticeable).
Global treatment assessment by participants | At the conclusion of the study, approximately 2 weeks later.
  On a scale from 0 to 10 (where 0 = no response or not satisfied at all, and 10 = excellent response or exceptionally satisfied) after the treatment. A score of ≥ 6 out of 10 will indicate responders.
Clinical assessment of the skin condition by a specialist. | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  Clinical assessment of the skin condition (localization of the vesicles, extent or lack thereof to the skin, observation of other related factors: fever, muscle pain, lymph node inflammation...).
Mild adverse events. | Through study completion, apprroximately 2 weeks.
  Evaluate the incidence of other mild and transient adverse events related to the product.
Mean duration of the episode | Through study completion, apprroximately 2 weeks
  Mean duration of the episode (MDE) due to cold sores (≤ 7 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Complutense Grupo Virtus, Alcalá de Henares, Madrid, Spain